CLINICAL TRIAL: NCT03923322
Title: Randomized Pilot Trial of Botanical Tincture for Symptoms of Irritable Bowel Syndrome Constipation Predominant (IBS-C) Diagnosed on ROME IV Criteria
Brief Title: Botanical Tincture for Symptoms of Irritable Bowel Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Budget limitations
Sponsor: Stamford Hospital (Other)
Responsible Party: Principal Investigator, Marc Brodsky, Director, Center for Integrative Medicine and Wellness, Stamford Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSH_Family Medicine_2018001
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Irritable Bowel Syndrome Characterized by Constipation

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Botanical Tincture (Experimental): The 12-week study includes a 2-week screening, 8-week treatment, and 2-week withdrawal periods. A 2-week screening period will be used to establish the presence and persistence of trial entry criteria and train patients in the mode of data collection. Participants randomly assigned to the Botanical Tincture arm at Week 2 will take 2.5 ml by mouth once a day at any time during the day that they choose. Participants who received Botanical Tincture during the study will be followed by a 2-week randomized withdrawal design to address the need for maintenance treatment to prevent sign or symptom recurrence. The participant will be randomly reassigned to receive either Botanical Tincture or placebo at a dosage of 2.5 ml once a day by mouth at any time during the day that they prefer.
  Interventions: Drug: Botanical Tincture
- Placebo (Placebo Comparator): Participants randomly assigned to placebo arm at Week 2 will take 2.5 ml by mouth once a day at any time during the day that they choose during the 8-week treatment period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Botanical Tincture — Study participants will meet with the Investigator at baseline and week 2, 6, and 10 after the study period begins. Trial continuation criteria at 2 weeks after the start of the study includes abdominal pain intensity and stool frequency. Participants randomized to Botanical Tincture will have a 2-week withdrawal period. On the visits study participants may expect to be asked about epidemiologic information, IBS medications, IBS Quality of Life survey instruments, and daily diary of pain scale, bloating scale, and number of bowel movements.
  Other Names: BT
  Arms: Botanical Tincture
Other: Placebo — Study participants will meet with the Investigator at baseline and week 2, 6, and 10 after the study period begins. Trial continuation criteria at 2 weeks after the start of the study includes abdominal pain intensity and stool frequency. On the visits study participants may expect to be asked about epidemiologic information, IBS medications, IBS Quality of Life survey instruments, and daily diary of pain scale, bloating scale, and number of bowel movements.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to investigate the feasibility of a follow-up larger RCT on the efficacy of Botanical Tincture to relieve abdominal pain in people with Irritable Bowel Syndrome Constipation Predominant (IBS-C).

DETAILED DESCRIPTION:
The randomized pilot trial will address subject recruitment, retention, and subject compliance with protocol. A secondary is to learn if people with IBS-C are able to tolerate Botanical Tincture and the effect of taking Botanical Tincture on abdominal pain, bloating, and bowel movements.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting ROME IV criteria for the diagnosis of irritable bowel syndrome that requires that patients have had recurrent abdominal pain on average at least 1 day per week during the previous 3 months that is associated with 2 or more of the following :
* Related to defecation (may be increased or unchanged by defecation)
* Associated with a change in stool frequency
* Associated with a change in stool form or appearance
* Abdominal Pain Intensity: average of worst daily (in past 24 hours) abdominal pain score of >= 3 on a 0 to 10 point scale over last week
* Stool Frequency: < or = to 3 Complete Spontaneous Bowel Movement(CSBM) in the previous week
* Reported bloating rating > or = 2 on 5-point scale [0 (absent) - 4 (very severe)] in previous week
* English speakers, as all surveys are in English

Exclusion Criteria:

* Patients with known hypersensitivity to any component of the trial drugs
* History of eating disorders
* Patients with a history of diseases with abdominal symptoms that can resemble IBS
* Presence of any other known acute or chronic gastrointestinal disorder
* History of abdominal surgery (cholecystectomy and appendectomy can be tolerated when performed at least one year previously)
* Pregnancy or breast feeding
* Current or past history of alcohol dependence
* Based on lack of adequate scientific evidence to predict drug-drug interaction in vivo, current use of strong inhibitors or inducers for CYP enzymes and participants are instructed not to take any medications that are strong inhibitors or inducers for CYP enzymes during the course of the study
* Vulnerable Subjects. The study will not include vulnerable subjects (such as, those with limited autonomy or those in subordinate hierarchical positions). Children, pregnant women, nursing home residents or other institutionalized persons, students, employees, fetuses, prisoners, and persons with decisional incapacity will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects recruited | 2 years
  60 subjects
Proportion of subjects who complete the study | 12 week study
  At least 80% subjects will complete study
Proportion of dosages of drug/placebo that are taken by participants | 12 week study
  At least 80% of dosages will be taken by participants

SECONDARY OUTCOMES:
Abdominal Pain Intensity: weekly average of worst daily (in past 24 hours) abdominal pain score scale of 0 (No pain) -10 (Worst imaginable pain) | 12 week study
  An Abdominal Pain Intensity Weekly Responder is defined as a patient who experiences a decrease in the weekly average of worst abdominal pain in the past 24 hours score (measured daily) of at least 30% compared with baseline weekly average.
Abdominal Bloating Intensity: weekly average of worst daily (in past 24 hours) abdominal bloating rating on a scale of 0 (absent) - 4 (very severe) | 12 week study
  A Bloating Intensity Weekly Responder is defined as a patient who experiences a decrease in the weekly average of worst bloating pain in the past 24 hours score (measured daily) of at least 30% compared with baseline weekly average
Bowel movement frequency: Number of Complete Spontaneous Bowel Movements (CSBMs) each week | 12 week study
  A Stool Frequency Weekly Responder is defined as a patient who experiences an increase of at least one CSBM per week from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Marc Brodsky, MD, Principal Investigator — Stamford Hospital
Locations (1):
- Stamford Health, Stamford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available from Marc Brodsky, MD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after publication for unlimited time
Access Criteria: Researcher